CLINICAL TRIAL: NCT07379840
Title: Post Marketing Surveillance for Finerenone Chronic Heart Failure in Korea
Brief Title: A Study to Learn More About How Safe Finerenone is and How Well it Works in Adults With Chronic Heart Failure in South Korea
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23041
Record Dates: First submitted 2025-12-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; Post-Marketing Surveillance
MeSH Terms: conditions — Heart Failure | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- finerenone group: Participants in Korea who are prescribed finerenone for treatment of chronic HF with left ventricular ejection fraction (LVEF) ≥40%.
  Interventions: Drug: finerenone (BAY94-8862)

INTERVENTIONS:
Drug: finerenone (BAY94-8862) — According to the prescription of the participating patient

SUMMARY:
This is an observational study in which data from people with chronic heart failure (HF) with left ventricular ejection fraction (LVEF) ≥ 40%. who will be receiving finerenone are studied.

The study is conducted to check the safety of finerenone after it is approved and available in South Korea.

Observational studies use data that are collected as part of routine medical care and participants do not receive any advice or any changes to healthcare as part of the study.

In this study, the data will be collected from participants who are receiving their usual treatment with finerenone as prescribed by their doctor according to the approved product information.

Heart failure with LVEF ≥ 40% is a condition which occurs when the left side of the heart does not pump blood out to the body as well as it should. Over time, the body does not get the amount of oxygen it needs. This can lead to shortness of breath and tiredness, making it difficult for people to do their daily tasks.

The study drug, finerenone, is already approved for doctors to prescribe to people with chronic heart failure. It works by blocking a specific receptor in the body called the mineralocorticoid receptor (MR). This helps reduce harmful effects in the heart, kidneys and blood vessels. Finerenone is different from older medicines in this group because it is more selective and may have fewer side effects, such as problems with the kidneys or high potassium levels in the blood.

The participants in this study will receive finerenone as prescribed independently by their doctors during routine practice according to the approved product information.

There have been studies in which researchers studied the effect and safety of finerenone in participants with chronic heart failure with LVEF ≥ 40%. These studies, however, included only a small number of South Korean participants. In this study, researchers will specifically gather data from South Korean participants to further understand the safety of finerenone.

The main purpose of this study is to learn more about how safe and effective finerenone is in adults with chronic heart failure with LVEF ≥ 40% in South Korea within approved local label when used in everyday medical practice.

To do this, researchers will collect any side effects or health problems that happen while patients are taking finerenone, and whether they are related to finerenone.

In addition, doctors will also look at how well finerenone works by measuring:

* Changes in investigator's treatment satisfaction with the treatment over time, including improvements in symptoms, quality of life and overall health status.
* Time to dose change of finerenone (for example, increasing the dose if needed).

Data will be collected from participants over one year after they enroll in the study or until they choose to leave the study. The data will come from participant's medical records or by interviewing the patient.

In this study, only available data from routine care will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 19 years or older
* With informed consent from subject or legal representative (Prioritizing patient consent)
* Finerenone naïve patients who are prescribed finerenone for treatment of chronic HF with LVEF ≥40%

Exclusion criteria:

* Contraindication according to the local label (including known hypersensitivity to the drug substance or any of its components)
* Patients participating in an investigational program with interventions outside of routine clinical practice (NYHA classes II-IV) in accordance with local label

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult chronic HF patients with LVEF ≥40% prescribed finerenone in routine clinical practice in Korea
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | 12 months from baseline
  including treatment emergent adverse events (TEAEs), adverse drug reactions (ADRs), unexpected AEs, unexpected ADRs, serious adverse events (SAEs), serious adverse drug reactions (SADRs), adverse events of special interest (AESI)

SECONDARY OUTCOMES:
Change from baseline in investigator's treatment satisfaction | at 1, 3, 6 and 12 months
  Investigator's treatment satisfaction will be assessed on a 7-point Likert-type scale ([1] Strongly agree; [2] Agree; [3] More or less agree; [4] Undecided; [5] More or less disagree; [6] Disagree; [7] Strongly disagree).
Time to dose change of finerenone | up to 12 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.

REFERENCES:
- See also: Click here for access to information about Bayer's transparency standards and Bayer studies. — https://clinicaltrials.bayer.com